CLINICAL TRIAL: NCT01546181
Title: Observational, Follow-up Study of Adaptive Optics Retinal Imaging in Controls and During Retinal or General Diseases
Brief Title: Retinal Imaging by Adaptive Optics in Healthy Eyes and During Retinal and General Diseases
Acronym: iPhot
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C10-03; 2010-A00492-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Retinal Dystrophies; Age-related Macular Degeneration; Arterial Hypertension; Diabetes; Traumatic Retinopathy; Toxic Retinopathies
Keywords: photoreceptors; retinal pigment epithelium; adaptive optics
MeSH Terms: conditions — Retinal Dystrophies; Macular Degeneration; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Controls: subjects older than 10 years old, with no know ocular or general disease
- Age-related macular degeneration
- inherited retinal dystrophies
- retinal trauma
- toxic retinopathies
- arterial hypertensive patients
- diabetic patients
- inflammatory diseases

SUMMARY:
Using an adaptive optics imaging device, retinal structures are observed in healthy and diseased subjects.

DETAILED DESCRIPTION:
Most cases of severe visual loss in developed countries are due to retinal diseases affecting a specialized class of neurons, the photoreceptors. Currently available systems for retinal imaging in humans do not allow neuronal imaging at the cellular level, which is crucial to understand, diagnose and monitor retinal diseases. In recent years, adaptive optics (AO) fundus imaging has proven its capability to image individual photoreceptor cells in the human retina. This technology is now reaching technical maturation. A prototypic AO system (manufactured by Imagine Eyes) is currently in operation in a clinical setting (Clinical Investigation Center 503) and has proven its reliability to monitor single photoreceptors over time. Yet, the clinical evaluation of AO imaging is still in its infancy, and biomarkers issued from AO imaging have not been validated. The goal of the iPhot project is thus to optimize the process of AO imaging (from the implementation of novel technical solution to image processing and data analysis) in order to obtain morphological, quantitative and longitudinal information concerning retinal microstructures in humans. For instance, we will aim at detecting early photoreceptor damage during retinal dystrophies.

ELIGIBILITY:
Inclusion Criteria:

* over 10 years old

Exclusion Criteria:

* ocular media opacities, unstable fixation

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: controls and patients with any kind of retinal alteration
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2010-10; Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
photoreceptor density | 01/12/2014
  the variations of the density of photoreceptors over time will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Michel Paques, MD, PhD, Principal Investigator — Quinze-Vingts Hospital, Paris
Locations (1):
- Clinical Investigation Center 503, Paris, France

REFERENCES:
- [Result] Paques M, Miloudi C, Kulcsar C, Leseigneur A, Chaumette C, Koch E. High-resolution imaging of gunn's dots. Retina. 2015 Jan;35(1):120-4. doi: 10.1097/IAE.0000000000000269. PMID 25077537
- [Result] Audo I, Gocho K, Rossant F, Mohand-Said S, Loquin K, Bloch I, Sahel JA, Paques M. Functional and high-resolution retinal imaging monitoring photoreceptor damage in acute macular neuroretinopathy. Graefes Arch Clin Exp Ophthalmol. 2016 May;254(5):855-64. doi: 10.1007/s00417-015-3136-6. Epub 2015 Sep 7. PMID 26344727
- [Result] Paques M, Brolly A, Benesty J, Lerme N, Koch E, Rossant F, Bloch I, Girmens JF. Venous Nicking Without Arteriovenous Contact: The Role of the Arteriolar Microenvironment in Arteriovenous Nickings. JAMA Ophthalmol. 2015 Aug;133(8):947-50. doi: 10.1001/jamaophthalmol.2015.1132. PMID 25997175
- [Result] Miloudi C, Rossant F, Bloch I, Chaumette C, Leseigneur A, Sahel JA, Meimon S, Mrejen S, Paques M. The Negative Cone Mosaic: A New Manifestation of the Optical Stiles-Crawford Effect in Normal Eyes. Invest Ophthalmol Vis Sci. 2015 Nov;56(12):7043-50. doi: 10.1167/iovs.15-17022. PMID 26523388
- [Result] Gocho K, Sarda V, Falah S, Sahel JA, Sennlaub F, Benchaboune M, Ullern M, Paques M. Adaptive optics imaging of geographic atrophy. Invest Ophthalmol Vis Sci. 2013 May 1;54(5):3673-80. doi: 10.1167/iovs.12-10672. PMID 23620431
- [Result] Koch E, Rosenbaum D, Brolly A, Sahel JA, Chaumet-Riffaud P, Girerd X, Rossant F, Paques M. Morphometric analysis of small arteries in the human retina using adaptive optics imaging: relationship with blood pressure and focal vascular changes. J Hypertens. 2014 Apr;32(4):890-8. doi: 10.1097/HJH.0000000000000095. PMID 24406779
- [Result] Errera MH, Coisy S, Fardeau C, Sahel JA, Kallel S, Westcott M, Bodaghi B, Paques M. Retinal vasculitis imaging by adaptive optics. Ophthalmology. 2014 Jun;121(6):1311-2.e2. doi: 10.1016/j.ophtha.2013.12.036. Epub 2014 Feb 25. No abstract available. PMID 24576889
- [Result] Faure C, Gocho K, Le Mer Y, Sahel JA, Paques M, Audo I. Functional and high resolution retinal imaging assessment in a case of ocular siderosis. Doc Ophthalmol. 2014 Feb;128(1):69-75. doi: 10.1007/s10633-013-9421-y. Epub 2013 Dec 13. PMID 24337723
- [Result] Bottin C, Grieve K, Rossant F, Pedinielli A, Mrejen S, Paques M. DIRECTIONAL VARIABILITY OF FUNDUS REFLECTANCE IN ACUTE MACULAR NEURORETINOPATHY: EVIDENCE FOR A CONTRIBUTION OF THE STILES-CRAWFORD EFFECT. Retin Cases Brief Rep. 2018 Fall;12 Suppl 1:S19-S24. doi: 10.1097/ICB.0000000000000701. PMID 29369084
- [Result] Jacob J, Paques M, Krivosic V, Dupas B, Couturier A, Kulcsar C, Tadayoni R, Massin P, Gaudric A. Meaning of visualizing retinal cone mosaic on adaptive optics images. Am J Ophthalmol. 2015 Jan;159(1):118-23.e1. doi: 10.1016/j.ajo.2014.09.043. Epub 2014 Oct 2. PMID 25284764
- [Result] Rosenbaum D, Mattina A, Koch E, Rossant F, Gallo A, Kachenoura N, Paques M, Redheuil A, Girerd X. Effects of age, blood pressure and antihypertensive treatments on retinal arterioles remodeling assessed by adaptive optics. J Hypertens. 2016 Jun;34(6):1115-22. doi: 10.1097/HJH.0000000000000894. PMID 27065002
- [Result] Rosenbaum D, Kachenoura N, Koch E, Paques M, Cluzel P, Redheuil A, Girerd X. Relationships between retinal arteriole anatomy and aortic geometry and function and peripheral resistance in hypertensives. Hypertens Res. 2016 Jul;39(7):536-42. doi: 10.1038/hr.2016.26. Epub 2016 Mar 24. PMID 27009576
- [Result] Faure C, Paques M, Audo I. Electrophysiological features and multimodal imaging in ritonavir-related maculopathy. Doc Ophthalmol. 2017 Dec;135(3):241-248. doi: 10.1007/s10633-017-9612-z. Epub 2017 Sep 12. PMID 28900746
- [Result] Boileve A, Jozwiak M, Malka D, Boige V, Le Roy F, Paques M, Ducreux M. Vision loss after chemotherapy: an irinotecan-induced retinopathy. Eur J Cancer. 2019 May;112:80-82. doi: 10.1016/j.ejca.2019.02.015. Epub 2019 Apr 1. No abstract available. PMID 30947025
- [Result] Paques M, Meimon S, Rossant F, Rosenbaum D, Mrejen S, Sennlaub F, Grieve K. Adaptive optics ophthalmoscopy: Application to age-related macular degeneration and vascular diseases. Prog Retin Eye Res. 2018 Sep;66:1-16. doi: 10.1016/j.preteyeres.2018.07.001. Epub 2018 Jul 17. PMID 30010022
- [Result] Sodi A, Germain DP, Bacherini D, Finocchio L, Pacini B, Marziali E, Lenzetti C, Tanini I, Koraichi F, Coriat C, Nencini P, Olivotto I, Virgili G, Rizzo S, Paques M. IN VIVO OBSERVATION OF RETINAL VASCULAR DEPOSITS USING ADAPTIVE OPTICS IMAGING IN FABRY DISEASE. Retina. 2020 Aug;40(8):1623-1629. doi: 10.1097/IAE.0000000000002648. PMID 31568064
- [Result] Errera MH, Laguarrigue M, Rossant F, Koch E, Chaumette C, Fardeau C, Westcott M, Sahel JA, Bodaghi B, Benesty J, Paques M. High-Resolution Imaging of Retinal Vasculitis by Flood Illumination Adaptive Optics Ophthalmoscopy: A Follow-up Study. Ocul Immunol Inflamm. 2020 Nov 16;28(8):1171-1180. doi: 10.1080/09273948.2019.1646773. Epub 2019 Oct 1. PMID 31573376
- [Result] Paques M, Rossant F, Finocchio L, Grieve K, Sahel JA, Pedinielli A, Mrejen S. ATTENUATION OUTER RETINAL BANDS ON OPTICAL COHERENCE TOMOGRAPHY FOLLOWING MACULAR EDEMA: A Possible Manifestation of Photoreceptor Misalignment. Retina. 2020 Nov;40(11):2232-2239. doi: 10.1097/IAE.0000000000002738. PMID 31922497
- [Result] Gallo A, Chaigneau E, Jublanc C, Rosenbaum D, Mattina A, Paques M, Rossant F, Girerd X, Leban M, Bruckert E. IGF-1 is an independent predictor of retinal arterioles remodeling in subjects with uncontrolled acromegaly. Eur J Endocrinol. 2020 Mar;182(3):375-383. doi: 10.1530/EJE-19-0390. PMID 31972545
- [Derived] Jacob J, Krivosic V, Paques M, Tadayoni R, Gaudric A. CONE DENSITY LOSS ON ADAPTIVE OPTICS IN EARLY MACULAR TELANGIECTASIA TYPE 2. Retina. 2016 Mar;36(3):545-51. doi: 10.1097/IAE.0000000000000737. PMID 26418443